CLINICAL TRIAL: NCT05715268
Title: Moving MS Bladder Dysfunction Into the 21st Century: Developing Novel and Accessible Ways to Treat Dysfunction in the Home - a Three Month Single Arm Open Label Feasibility Pilot With Waitlist Control
Brief Title: Wearables for the Bladder: an In-home Treatment Feasibility Pilot Study
Acronym: WeB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A137172
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis; Urinary Bladder, Overactive
Keywords: multiple sclerosis; remote; wearables; overactive bladder; pelvic floor physical therapy
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Three month feasibility pilot with a standard of care control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- WeB and pelvic floor physical therapy group (Experimental): This group will receive standard PFPT as well as WeB device for 12 weeks, and MS-symptom (including bladder bother) related questionnaires at baseline, 12 weeks and 6 months post intervention. Participants will also be provided with a remote activity monitor to use during the study.
  Interventions: Device: WeB; Other: Standard pelvic floor physical therapy
- Control pelvic floor physical therapy group (Active Comparator): This group will receive standard PFPT for 12 weeks. MS-symptom (including bladder bother) related questionnaires at baseline, 12 weeks and 6 months after the last PFPT visit.
  Patients will be invited to use WeB devices after this time.
  Interventions: Other: Standard pelvic floor physical therapy

INTERVENTIONS:
Device: WeB — Participants will be given WeB devices and trained on the use of these devices for home therapy, including the associated mobile applications. Participants will be given home programs and given a schedule to use the WeB devices at home on their own time. At their standard visit participants will have their WeB device use checked and progressed as the therapist deems appropriate.
  An in-person visit will be scheduled to re-evaluated participants at the 12 week study completion.
  Arms: WeB and pelvic floor physical therapy group
Other: Standard pelvic floor physical therapy — Baseline will consist of a standard PFPT evaluation. Regular visits (tele-video visits or in-person depending on the patients preference) will be scheduled every week for the first 4 weeks and then every other week at the discretion of the therapist. A total of 8-10 visits will be scheduled over the 12 weeks of the study. Participants will be given home exercise programs (as per standard PFPT).
  An in-person visit will be scheduled to re-evaluated participants at the 12 week study completion.

SUMMARY:
The goal is to investigate the feasibility and effects of adding "wearables for the bladder" devices to conventional pelvic floor physical therapy (PFPT) to bladder function, in people with multiple sclerosis (MS).

DETAILED DESCRIPTION:
The participants baseline pelvic floor and bladder function will be assessed by a pelvic floor physical therapist as per standard care, and online MS-symptom questionnaires (i.e., quality of life, bladder bother/symptoms, falls, fatigue, depression). Participants will be trained on the maintenance and use of "wearable for the bladder" (WeB) devices. Participants will receive standard PFPT intervention care, and will be asked to further train using the WeB devices. 8-10 sessions will be conducted over telehealth or in person as per standard protocol. At 12 weeks, participants will return to clinic for pelvic floor and bladder function assessment.

A control group will receive standard PFPT intervention care as well as online MS-symptom questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis
* Assigned Female at birth and whose sex is currently Female
* Mild/moderate bladder dysfunction (bowel/bladder functional systems scores = 0-2 or Bladder control scale >0)
* California residents
* Wifi in the home and personal smartphone (using Apple operating system)
* Able to walk with or without assistive device
* Manual muscle test score of 2 or more.

Exclusion Criteria:

* Undergone treatment for bladder dysfunction symptoms within 3 months
* Current urinary tract infection
* Recent (~30 days) relapse
* Any cognitive, dexterity or visual impairment so severe that it precludes use of the wearables for the bladder tool or ability to use a smartphone
* Pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Net Promoter Score | 12 weeks
  This is a response to a single question: "How likely would you be to recommend [participation in a study or treatment like this] to a friend or family member with Multiple Sclerosis?" Net promoter scores range from 0 (would not recommend) to 10 (would definitely recommend).
Health Information Technology Usability Evaluation Scale (Health-ITUES) - Ease of use | 12 weeks
  In response to four statements about the ease of use for the wearables for the bladder (WeB): ranking each from 1 (strongly disagree) to 5 (strongly agree). Scores range from 5-20. Lower scores relate to less ease of use.
Health Information Technology Usability Evaluation Scale (Health-ITUES) - Perceived usefulness | 12 weeks
  In response to nine statements about the Perceived usefulness of the wearables for the bladder (WeB) ranking each from 1 (strongly disagree) to 5 (strongly agree). Scores range from 5-20. Lower scores relate to less perceived usefulness.
System usability scale | 12 weeks
  It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree (5) to Strongly disagree (1) - ranking each from 1 (strongly disagree) to 5 (strongly agree). Scores range from 10-100. Lower scores relate to less usability.
Adherence as measured by percent usage | 12 weeks
  Usage ranges from 0-100% use, where 100% use would be total adherence to prescribed use duration.

SECONDARY OUTCOMES:
Change in Overactive bladder symptom scale; OABSS | Baseline and 12 weeks
  The questionnaire consists of 4 questions on overactive bladder symptoms with maximum scores ranging from 2 to 5: daytime frequency (2 points), night-time frequency (3 points), urgency (5 points), and urge urinary incontinence (5 points). The total score ranges from 0 to 15 points, with higher scores indicating higher symptom severity.
Change in Overactive bladder symptom scale; OABSS | Baseline and 9 months
  The questionnaire consists of 4 questions on overactive bladder symptoms with maximum scores ranging from 2 to 5: daytime frequency (2 points), night-time frequency (3 points), urgency (5 points), and urge urinary incontinence (5 points). The total score ranges from 0 to 15 points, with higher scores indicating higher symptom severity.
Change in the number of daily leakage episodes | Baseline and 12 weeks
  Change in number of leaks per day as measured by the wearables for the bladder application. The patient will manually enter the number of leaks into the application.
Change in the number of daily leakage episodes | Baseline and 9 months
  Change in number of leaks per day as measured by the wearables for the bladder application. The patient will manually enter the number of leaks into the application.
Change in the frequency of daily voiding episodes | Baseline and 12 weeks
  Change in the frequency of voids per day as measured by the wearables for the bladder application. The patient will manually enter voids into the application.
Change in the frequency of daily voiding episodes | Baseline and 9 months
  Change in the frequency of voids per day as measured by the wearables for the bladder application. The patient will manually enter voids into the application.
Change in the 29 item- multiple sclerosis quality of life survey (MSQOL-29) | Baseline and 12 weeks
  Measurement of changes in quality of life via the MSQOL-29: consists of seven multi-item subscales: 'physical function' (six items); 'sexual function' (four items); 'bodily pain', 'emotional well-being', 'energy', 'cognitive function' and 'health distress' (three items); and four single-item subscales ('social function', 'health perceptions', 'overall quality of life', and 'change in health') which form two composite scores (Physical Health Composite, (PHC) and Mental Health Composite, (MHC))
Change in the SymptoMScreen survey | Baseline and 9 months
  Measurement of changes in quality of life via the SymptoMScreen - a 12 question survey asking about MS symptoms affecting everyday life. Each question is graded on a scale of 0 - not affected at all, to 6 - Total limitation. Scores are summed and range from 0 -72.
Satisfaction with using WeB devices | 12 weeks
  Using a single question ("Do you like this tool?") graded on a Likert scale (0, do not like at all, 100, like very much). Higher scores indicate higher satisfaction.

OTHER OUTCOMES:
Change in average quality of sleep | baseline, and 12 weeks
  Remote monitoring devices will provide passive sleep scores rated as a percentage. Higher percentages reflect better sleep scores.
Change in average daily step count | baseline, and 12 weeks
  Remote monitoring devices will provide passive daily step count as a number above 0- the daily step counts over the study will be averaged. Higher steps reflect more physical activity.
Change in Heart rate variability | baseline, and 12 weeks
  Remote monitoring devices will provide passive heart rate variability (in milliseconds) - heart rate variability is the variation in the time between heartbeats, and lowering heart rate variability may indicate an increase in stress or strain.
Change in Bladder control scale; BLCS | Baseline and 12 weeks
  Four-item instrument assessing the extent to which bladder problems have an impact on everyday activities over the last 4 weeks.
  Raw scores are summed to create a total score ranging from 0 to 22 (higher scores indicate more severe bladder bother)
Change in application pelvic fitness test; control | Baseline and 12 weeks
  Change in pelvic floor muscle control - graded from 0-50
Change in application pelvic fitness test; speed | Baseline and 12 weeks
  Change in pelvic floor muscle contraction speed - graded from 0-10
Change in application pelvic fitness test; endurance | Baseline and 12 weeks
  Change in pelvic floor muscle endurance - graded from 0-20

CONTACTS AND LOCATIONS:
Overall Officials: Valerie J Block, DPTSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, Weill Institute for Neurosciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No